CLINICAL TRIAL: NCT00738257
Title: A 2 Year Prospective, Multicentre, Open-label, Randomised, Controlled Study to Investigate the Effectiveness of Pamidronate in the Prevention of Bone Loss in de Novo Renal Transplant Patients (With a PTH > 150pg/ml) on a Ciclosporin A and Glucocorticoid Based Immunosuppressive Regimen.
Brief Title: A Prospective, Multicentre, Open-label Randomised Controlled Study to Investigate the Effectiveness of Pamidronate in the Prevention of Bone Loss in de Novo Renal Transplant Patients.
Acronym: SMART
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEO-GB-50; ARE-GB-01
Record Dates: First submitted 2008-08-18; First posted 2008-08-20 (Estimated); Last update posted 2010-05-17 (Estimated); Status verified 2010-05

CONDITIONS: Bone Loss
Keywords: Renal; transplant,; pamidronate,; ciclosporin,; Ciclosporin A,; steroids,; bone mineral density,; fracture rates; immunosuppressive; regimen
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Pamidronate

ARMS (1):
- Parmidronate (Experimental)
  Interventions: Drug: Pamidronate

INTERVENTIONS:
Drug: Pamidronate

SUMMARY:
The purpose of the study was to evaluate the effect of Pamidronate on bone mineral density loss and fracture rates up to 2 years, in post renal-transplant subjects on a Ciclosporin A and glucocorticoid based immunosuppressive regimen.

ELIGIBILITY:
Inclusion Criteria:

1. First or second kidney transplant recipients, aged 18-75 years, PTH > 150 pg/ml
2. De novo patients scheduled to receive ciclosporin A and prednisolone based immunosuppression.

Exclusion Criteria:

1. Previous or current bone disease unrelated to end stage renal failure.
2. Patients with PTH < 150pg/ml who may be at risk of adynamic bone disease.
3. Treatment at any time with a bisphosphonate.
4. d. Calcitonin treatment during the previous month.
5. Malignancy (current or history within last 5 years)
6. Pregnancy or lactation, or women of childbearing potential unwilling to use an effective form of contraception for the 12 month duration of the study.

Protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2000-06; Primary Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Cunningham, MD, Principal Investigator — Royal London Hospital
Locations (1):
- Novartis Investigative Site, Frimley, United Kingdom

REFERENCES:
- [Derived] Walsh SB, Altmann P, Pattison J, Wilkie M, Yaqoob MM, Dudley C, Cockwell P, Sweny P, Banks LM, Hall-Craggs M, Noonan K, Andrews C, Cunningham J. Effect of pamidronate on bone loss after kidney transplantation: a randomized trial. Am J Kidney Dis. 2009 May;53(5):856-65. doi: 10.1053/j.ajkd.2008.11.036. PMID 19393473